CLINICAL TRIAL: NCT01541930
Title: An Open, Uncontrolled Study Investigating the Safety and Efficacy of GK567 in the Deodorization of Malodorous Infected Cutaneous Fungating Neoplastic Tumours, Over 14 Days of Treatment
Brief Title: An Open, Uncontrolled Study of GK567 in the Deodorization of Malodorous Fungating Neoplastic Tumours
Acronym: GK567
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDT.07.SPR.27013
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-01

CONDITIONS: Malodorous Infected Cutaneous Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GK567 (Experimental): GK567: Metronidazole Gel 0.75% Once or twice daily, for 14 days, up to 30g
  Interventions: Drug: GK567

INTERVENTIONS:
Drug: GK567 — Once or twice daily, for 14 days, up to 30 g per day
  Other Names: GK567: Metronidazole Gel 0.75%

SUMMARY:
This clinical trial objective is to investigate the safety and efficacy of GK567 to alleviate malodour of foul smelling, anaerobically infected fungating neoplastic tumours, over 14 days of treatment.

The clinical hypothesis is that the success rate is no worse than 70% in the population of interest, where success for a patient is defined as a smell score of 0 or 1 at Day 14/end of treatment, as assessed by the Study Investigator.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a male or female aged between 20 years or older.
* The subject has a cutaneous fungating neoplastic tumour with a smell that suggests established or early infection, with a minimum score of 2 (i.e. mildly offensive smell) on a 0-4 smell scale, (based on the Study investigator's assessment)

Exclusion Criteria:

* The subject is currently receiving systemic antibiotics or received in the last 2 weeks,
* The subject is currently receiving systemic or topical Metronidazole or received in the last week,
* The subject is currently receiving topical antibiotics or received such treatment applied on cutaneous fungating neoplastic tumour in the last 1 week,
* The subject already receives any topical treatment on the cutaneous fungating neoplastic tumour

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Galderma investigational site, Kanagawa
  - Galderma investigational site, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: April 2012 to December 2012 in Japan
Groups:
- GK567: Metronidazole Gel 0.75%, Once or twice daily, for 14 days, up to 30g
Period: Overall Study
Arm/Group | GK567
Started | 21
Completed | 20
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All patients who received the treatment at least once (Safety population) were included in all efficacy and safety analyses.
Arm/Group | GK567
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Region of Enrollment [Number; unit: participants]
  Japan | 21
Primary Disease [Number; unit: participants]
  Breast Cancer | 21
  Other Cancer | 0
Skin Ulcer Size [Mean (Standard Deviation); unit: cm^2] | 68.6 (35.4)

OUTCOME MEASURES:

1. Primary Outcome: The Success Rate
Description: The success rate, where success for a patient is defined as a smell score of 0 or 1 (0: No smell, 1: Smell present but not offensive) as assessed by the Study Investigator
Time Frame: at Day 14 (end of treatment)
Population: All patients who received the treatment at least once (Safety population) were included in all efficacy and safety analyses. Only observed cases were part of the analyses. If the primary endpoint was missing, an additional analysis of this endpoint was performed using the last observation carried forward (LOCF) to impute the missing data.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | GK567
Number analyzed (Participants) | 21
percentage of participants | 95.2 [79.3 to 99.8]

2. Secondary Outcome: Smell Score by Investigator
Description: Tumour smell score was evaluated by the Study Investigator using the following scale; 0: No smell, 1: Smell present but not offensive, 2: Mildly offensive smell, 3: Moderately offensive smell, 4: Extremely offensive smell
Time Frame: on Days 0 (baseline), 7, and 14
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- GK567, Day 0: Metronidazole Gel 0.75%, Tumour smell score evaluated on Day 0 (Baseline)
- GK567, Day 7: Metronidazole Gel 0.75%, Tumour smell score evaluated on Day 7
- GK567, Day 14: Metronidazole Gel 0.75%, Tumour smell score evaluated on Day 14. One patient was withdrawn on Day 7 due to subject's request.
Arm/Group | GK567, Day 0 | GK567, Day 7 | GK567, Day 14
Number analyzed (Participants) | 21 | 21 | 20
participants
  0: No smell | 0 | 11 | 13
  1: Smell present but not offensive | 0 | 5 | 6
  2: Mildly offensive smell | 13 | 2 | 0
  3: Moderately offensive smell | 3 | 3 | 1
  4: Extremely offensive smell | 5 | 0 | 0

3. Secondary Outcome: Smell Score by Nurse
Description: Tumour smell score was evaluated by the Nurse using the following scale; 0: No smell, 1: Smell present but not offensive, 2: Mildly offensive smell,3: Moderately offensive smell, 4: Extremely offensive smell
Time Frame: on Days 0 (baseline), 7, and 14
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- GK567, Day 14: Metronidazole Gel 0.75%, Tumour smell score evaluated on Day 14. One patient was withdrawn on Day 7 by Subject's request.
Arm/Group | GK567, Day 0 | GK567, Day 7 | GK567, Day 14
Number analyzed (Participants) | 21 | 21 | 20
participants
  0: No smell | 1 | 12 | 15
  1: Smell present but not offensive | 3 | 4 | 4
  2: Mildly offensive smell | 9 | 2 | 1
  3: Moderately offensive smell | 3 | 2 | 0
  4: Extremely offensive smell | 5 | 1 | 0

4. Secondary Outcome: Smell Score by Patient
Description: Tumour smell score was evaluated by the Patient using the following scale; 0: No smell, 1: Smell present but not offensive, 2: Mildly offensive smell,3: Moderately offensive smell, 4: Extremely offensive smell
Time Frame: on Days 0 (baseline), 7, and 14
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | GK567, Day 0 | GK567, Day 7 | GK567, Day 14
Number analyzed (Participants) | 21 | 21 | 20
participants
  0: No smell | 1 | 9 | 16
  1: Smell present but not offensive | 8 | 12 | 4
  2: Mildly offensive smell | 6 | 0 | 0
  3: Moderately offensive smell | 4 | 0 | 0
  4: Extremely offensive smell | 2 | 0 | 0

5. Secondary Outcome: Appearance (Volume and Nature of Discharge at Cutaneous Ulcer)
Description: Appearance score was evaluated by the Study Investigator using the following scale; 0: None (No discharge, e.g. frequency of dressing change: once daily), 1: Mild (Dressing need to be Changed twice daily), 2: Moderate (Dressing need to be Changed 3 times daily), 3: Marked (Dressing need to be Changed >3 times daily / Bloody).
Time Frame: on Days 0 (baseline), 7, and 14
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- GK567, Day 0: Metronidazole Gel 0.75%, Appearance score evaluated on Day 0 (baseline)
- GK567, Day 7: Metronidazole Gel 0.75%, Appearance score evaluated on Day 7
- GK567, Day 14: Metronidazole Gel 0.75%, Appearance score evaluated on Day 14. One patient was withdrawn on Day 7 by Subject's request.
Arm/Group | GK567, Day 0 | GK567, Day 7 | GK567, Day 14
Number analyzed (Participants) | 21 | 21 | 20
participants
  0 None | 1 | 5 | 7
  1 Mild | 12 | 12 | 10
  2 Moderate | 3 | 0 | 1
  3 Marked | 5 | 4 | 2

6. Secondary Outcome: Pain (Visual Analogue Scale)
Description: The pain linked to the fungating tumour over the last 24 hours was evaluated by the patient. The pain was graded using a 100 mm linear visual analogical scale (graded from 0 mm = no pain to 100 mm = severe pain).
Time Frame: on Days 0 (baseline), 7, and 14
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm
Groups:
- GK567, Day 0: Metronidazole Gel 0.75%, Pain evaluation on Day 0 (baseline) by Visual Analogue Scale (mm)
- GK567, Day 7: Metronidazole Gel 0.75%, Pain evaluation on Day 7 by Visual Analogue Scale (mm)
- GK567, Day 14: Metronidazole Gel 0.75%, Pain evaluation on Day 14 by Visual Analogue Scale (mm) One patient was withdrawn on Day 7 by Subject's request
Arm/Group | GK567, Day 0 | GK567, Day 7 | GK567, Day 14
Number analyzed (Participants) | 21 | 21 | 20
mm | 28.3 (29.1) | 25.9 (27.1) | 22.2 (25.3)

ADVERSE EVENTS:
Time Frame: Overall study, 14 days (treatment period)
Groups:
- GK567: Metronidazole Gel 0.75%, Once or twice daily, for 14 days, up to 30 g
Arm/Group | GK567
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 14/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GK567 (N=21)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GK567 (N=21)
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Somnolence (Nervous system disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No